### **Research Study Informed Consent Document**

**Study Title for Participants:** Testing the addition of a new immunotherapy drug, Atezolizumab (MPDL3280A), to the usual chemoradiation (CRT) therapy treatment for Limited Stage Small Cell Lung Cancer (LS-SCLC)

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: NRG-LU005, Limited Stage Small Cell Lung Cancer (LS-SCLC): A Phase III Randomized Study of Chemoradiation Versus Chemoradiation Plus Atezolizumab (MPDL3280A) (NCT03811002) (02-JUNE-2021)

## **Overview and Key Information**

## What am I being asked to do?

We are asking you to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this research study because you have limited-stage small cell lung cancer that has not spread outside your chest.

## Taking part in this study is your choice.

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.

## Why is this study being done?

This study is being done to answer the following question: Can we lower the chance of small cell lung cancer growing or spreading by adding an immunotherapy drug (atezolizumab) to the usual treatment for this type of cancer?

We are doing this study to find out if this approach is better or worse than the usual approach for your type of cancer. The usual approach is defined as care most people get for small cell lung cancer.

# What is the usual approach to my limited stage small cell lung cancer? (18-SEPT-2020)

The usual approach for patients with limited-stage small cell lung cancer who are not in a study is treatment with chemotherapy and radiation therapy. Some patients also receive low dose radiation to the brain to decrease the chance of the cancer spreading to the brain. The five year survival rate for patients who get the usual approach for this cancer is about 25-30% (or 25-30 patients out of 100).

## What are my choices if I decide not to take part in this study?

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.
- You may choose not to be treated for cancer.
- You may choose to only get comfort care to help relieve your symptoms and not get treated for your cancer.

## What will happen if I decide to take part in this study? (18-SEPT-2020)

If you decide to take part in this study, you will receive chemotherapy (etoposide along with cisplatin or carboplatin) and radiation (called chemoradiation therapy or CRT) for up to 7 weeks, or you will get usual CRT for up to 7 weeks plus the study drug, atezolizumab, for up to one year or until your cancer gets worse or the side effects become too severe. If you are able to receive brain radiation, you will receive it after you complete CRT.

You will be monitored for side effects during treatment. After you finish your study treatment, your doctor will still watch you for side effects. During the first 2 years after treatment, your doctor will check you every 3 months. During year 3, they will check you every 6 months, then annually unless your doctor thinks you need to be seen sooner.

## What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.

#### **Risks**

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that the CRT plus atezolizumab may not be as good as CRT at shrinking your cancer and keeping your cancer from coming back.

There is also a risk that you could have side effects from the atezolizumab. These side effects may be worse and may be different than you would get with the usual approach for your cancer.

Some of the most common side effects of atezolizumab that the study doctors know about are:

- Lung inflammation
- Liver inflammation
- Diarrhea
- Abdominal pain/tenderness
- Hormone gland problems (pituitary, thyroid, adrenal glands and pancreas)
- Inflammation of the eye
- Nervous system problems such as weakness, numbness/tingling in hands and feet, confusion, changes in mood

There may be some risks that the study doctors do not yet know about.

#### **Benefits**

There is evidence that adding the study drug, atezolizumab, to CRT is effective in shrinking a different type of lung cancer (non-small cell lung cancer). It is unknown if atezolizumab is effective in small cell lung cancer. It is not possible to know now if the atezolizumab will extend your life or extend your time without cancer compared to the usual approach. This study will help the study doctors learn things that will help people in the future.

## If I decide to take part in this study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible because it is important that you stop safely. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

## Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes and the study is no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.
- You do not follow the study rules.
- For women: You become pregnant while on the study.
- The study is stopped by the National Cancer Institute (NCI), Institutional Review Board (IRB), Food and Drug Administration (FDA), or NRG Oncology. The study sponsor is the organization who oversees the study.

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or member of the research team.

## What is the purpose of this study? (03-AUG-2022)

The purpose of this study is to compare the usual treatment to atezolizumab plus the usual treatment. The addition of the study drug, atezolizumab, to the usual treatment could shrink your cancer and prevent it from returning. But, it could also cause side effects, which are described in the risks section below.

This study will help the study doctors find out if this different approach is better, the same or worse than the usual approach. To decide if it is better, the study doctors will be looking to see if the study drug increases the average lifespan of patients by 6 months or more compared to the usual approach.

This immunotherapy drug, atezolizumab, is approved by the FDA for use in metastatic non-small cell lung cancer for patients whose cancer progresses. It is now approved by the FDA for use in metastatic small cell lung cancer. But, it is not approved for use in limited stage small cell lung cancer.

There will be about 545 people taking part in this study.

## What are the study groups? (03-AUG-2022)

This study has 2 study groups. All participants will have received one cycle of chemotherapy before entering the study. On the study all participants will receive 3 cycles of chemotherapy (for a total of 4 cycles including the one cycle of chemotherapy received before entering the study), plus radiation. If your study doctor wants you to receive brain radiation, you will receive it after you complete chemotherapy and radiation (CRT).

#### • Group 1

If you are in this group, you will get the usual chemotherapy used to treat this type of cancer (etoposide and either cisplatin or carboplatin) three days in a row through a vein (intravenously) every 3 weeks for 3 cycles; each cycle equals 21 days. The etoposide will be given on days 1-3 of each cycle, the cisplatin or carboplatin on day 1 of each cycle. In addition, you will receive the usual radiation to your tumor. Radiation will be given either twice a day for approximately 3 weeks or once a day for approximately 6-7 weeks.

There will be about 272 people in this group.

## • Group 2

If you are in this group, you will get the same chemotherapy and radiation as noted above, plus the study drug called atezolizumab. The atezolizumab will be given through a vein in your arm on days 1 or 2 of each chemotherapy cycle and will continue every 3 weeks for up to one year or until your disease gets worse or the side effects become too severe.

There will be about 273 people in this group.

We will use a computer to assign you to one of the study groups. This process is called "randomization." It means that your doctor will not choose and you cannot choose which study group you are in. You will be put into a group by chance. You will have equal chance of being in Group 1 or Group 2.

Another way to find out what will happen to you during this study is to read the chart below. Start reading at the left and reach across to the right, following the lines and arrows.



## What exams, tests, and procedures are involved in this study? (22-FEB-2021)

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if it is safe for you to take part in the study. In addition to the usual care you could get even if you were not in a study, you will need a blood test to check for the hepatitis virus if you have not previously been tested.

If you join the study, you will have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Listed below are exams, tests, and procedures that need to be done as part of this study to monitor your safety and health, but may not be included in the usual care. We will use them to carefully follow the effects of the study treatment, including preventing and managing side effects.

• A blood test to monitor your thyroid function (Group 2 participants only)

This study will use genetic tests that may identify changes in the genes in your body's cells, specifically in the cancer cells. Your genes carry information about you and your family, from the color of your eyes to health conditions for which you may be at risk, such as certain kinds of cancer.

Some exams, tests, and procedures are a necessary part of the research study, but would not be included in usual care. Listed below are procedures that will be done for research purposes only.

#### Tissue Sample

Your study doctor will need to use some of the tissue leftover from your biopsy when you were diagnosed with cancer. This sample is a required part of the study and will be used to confirm your diagnosis of small cell lung cancer and also to test your cancer cells for the presence of markers that may help the immune system fight cancer. If any of the tissue is leftover and you choose to give your consent, it will be stored for biobanking. Biobanking will be discussed in the section on optional studies.

#### **Blood Samples**

You will need to give blood samples for studies that test for the presence of marker that may be related to the immune system's ability to fight cancer. You will need to give blood before you start treatment. You and your study doctor will not get the results of this testing.

You also will have an opportunity to participate in optional research that uses your tissue and blood specimens. There is more information about this part of the study at the end of the consent form.

#### Symptoms Survey

If you speak English, Spanish, French or Japanese, you will be asked to answer questions about your symptoms and side effects of treatment. Researchers will use this information to learn more about how cancer and cancer treatment affects people.

You will be asked to fill out these forms at the following times, and each time it will take about 5 to 10 minutes to complete:

- After registration but within 7 days before you start CRT treatment (protocol cycle 1);
- During CRT treatment (days 8 and 15 of protocol cycle 1-3 of chemotherapy)
- At the end of CRT, 6 months after CRT, and 15 months after completion of CRT.

Since this is a research survey, the responses you provide will not be shared with your doctor. If you are having any severe symptoms, health issues or other concerns, please be sure to discuss these with your doctor or nurse right away.

At the end of the study, the answers you provided will be used to learn more about how cancer and cancer treatment affects patients, and it may help future patients.

#### Quality of Life Study

If you speak English, Spanish, French or Japanese and choose to take part in this study, you will be asked to answer questions about physical and emotional well-being and fatigue. Researchers will use this information to understand how atezolizumab impacts side effects and quality of life after treatment.

You will be asked to fill out these forms at the following times, and each time it will take about 5 to 10 minutes to complete:

- After registration but within 7 days before you start CRT treatment (protocol cycle 1);
- At the end of CRT, 3, 6, 15, and 21 months after CRT, and then every other year for up to 5 years after the end of treatment.

Since these forms are being used for research, the responses you provide will not be shared with your study doctor. If you have any serious health issues or other concerns, please talk with your doctor or nurse right away.

## Option for completing Symptoms Survey and Quality of Life with a personal electronic device

If you speak English or Spanish, after completing the first set of questions described above, you will have the option of completing the rest of the survey by paper or by an electronic device (not available for patients who read Japanese or French only). If you choose to complete the survey with an electronic device, you will enter your answers to the survey via a personal electronic device such as your smart phone or tablet. This may result in minor increases in your cell phone data usage. In some cases, your clinic may provide a tablet for you to answer the survey during your clinic visits. Whether you use a personal device or a tablet supplied by the clinic, your answers and personal information will not be stored on the device. Your answers will be sent to the research database and will be kept private in the same way listed in the later section about who will see your medical records. Your e-mail address will only be used for this survey study and will not be used for mail or marketing purposes. NRG Oncology will not keep your e-mail address. All patients will complete the survey before treatment on paper. After that, you can choose to complete questionnaires using an electronic device, see Appendix I of this document for more information.

#### Please circle your answer:

I choose to use the electronic software for completing the Symptom Survey and Quality of Life forms. I agree to fill out the Symptoms Survey and Quality of Life forms electronically (after treatment has started).

YES NO

## What risks can I expect from taking part in this study? (19-DEC-2023)

#### **General Risks**

If you choose to take part in this study, there is a risk that the CRT plus atezolizumab may not be as good as the usual approach for your cancer at shrinking or stabilizing your cancer and preventing it from coming back.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The treatments used in this study could be very harmful to an unborn or newborn baby. There may be some risks that doctors do not yet know about. For women who can become pregnant, it is very important that you check with your study doctor about what types of birth control or

pregnancy prevention to use during the study and for 5 months (150 days) after the last dose of atezolizumab.

This study will use a sample of your tissue. Generally, your hospital will keep some of your tissue. This tissue may be used to help treat your cancer in the future. Because this study will need to use some of this tissue, there is a small risk that it could be used up.

#### **Genetic Testing Risks**

The genetic tests used in this study will examine your blood samples for genetic traits that can mean better response to atezolizumab than other people who don't have the same genetic traits as you. This change also may be passed down through your family. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down.

Genetic tests can reveal information about you and also about your relatives. Finding these changes would not affect your treatment in this study. However, they could affect your health in other ways. If there are changes found that could cause health problems, your study doctor will talk with you about what further genetic testing may mean for you and your family. He or she also may suggest that you talk with a genetics counselor to learn more. You or your insurance plan would have to pay for any genetic tests and visits to a genetic counselor done outside of this study.

#### **Side Effect Risks**

The radiation therapy, chemotherapy and immunotherapy used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and let you know if changes occur that may affect your health. Most of these possible side effects could occur with the usual treatments or with the study treatment including atezolizumab. The most common risks related to drawing blood from your arm are brief pain and possibly a bruise.

There is also a risk that you could have other side effects from the study treatment.

Here are important things to know about side effects:

- 1. The study doctors do not know who will or will not have side effects.
- 2. Some side effects may go away soon, some may last a long time, and some may never go away.
- 3. Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.

• Your study doctor may adjust the usual treatments and the study drugs to try to reduce side effects.

This study is looking at a combination of the usual drugs used to treat this type of cancer plus a study drug (atezolizumab). This different combination of drugs may increase your side effects or may cause new side effects.

#### **Drug Risks**

The tables below show the most common and most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

Study Group 1 and Group 2 – Possible side effects of cisplatin and etoposide or carboplatin and etoposide are listed in the tables below. These drugs are part of the usual approach for treating this type of cancer:

#### Possible Side Effects of Cisplatin (Table Version Date: December 2, 2022)

### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Cisplatin, more than 20 and up to 100 may have:

- Infection, especially when white blood cell count is low
- Bruising, bleeding
- Anemia which may cause tiredness, or may require blood transfusions
- Kidney damage which may cause swelling, may require dialysis
- Hearing loss including ringing in the ears
- Nausea, vomiting
- Confusion
- Numbness, pain and tingling of the fingers, toes, arms and/or legs, loss of balance

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Cisplatin, from 4 to 20 may have:

- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Diarrhea
- Muscle weakness
- Change in taste
- Hair loss

#### RARE, AND SERIOUS

In 100 people receiving Cisplatin, 3 or fewer may have:

- Brain damage, Posterior Reversible Encephalopathy syndrome, which may cause headache, seizure, blindness
- Blood clot in lung which may cause swelling, pain, shortness of breath
- Seizure
- A new cancer, including leukemia, resulting from treatment of a prior cancer

#### Possible Side Effects of Etoposide (Table Version Date: December 3, 2021)

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Etoposide, more than 20 and up to 100 may have:

- Infection, especially when white blood cell count is low
- Bruising, bleeding
- Anemia which may cause tiredness, or may require blood transfusions
- Nausea, vomiting
- Sores in mouth which may cause difficulty swallowing
- Hair loss

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Etoposide, from 4 to 20 may have:

• Diarrhea, loss of appetite

#### RARE, AND SERIOUS

In 100 people receiving Etoposide, 3 or fewer may have:

- Liver damage which may cause yellowing of eyes and skin, swelling
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Blurred vision with chance of blindness
- A new cancer (including leukemia) resulting from treatment of a prior cancer
- Stevens-Johnson syndrome which may cause severe skin rash with blisters and peeling which can involve mouth and other parts of the body

#### Possible Side Effects of Carboplatin (Table Version Date: October 18, 2021)

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Carboplatin, more than 20 and up to 100 may have:

- Infection, especially when white blood cell count is low
- Bruising, bleeding

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Carboplatin, more than 20 and up to 100 may have:

- Anemia which may cause tiredness, or may require blood transfusions
- Vomiting, nausea
- Hair loss

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Carboplatin, from 4 to 20 may have:

- Diarrhea, constipation, belly pain
- Changes in taste
- Numbness and tingling in fingers and toes
- Weakness
- Swelling, redness, and pain at the site of the medication injection

#### RARE, AND SERIOUS

In 100 people receiving Carboplatin, 3 or fewer may have:

- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Visual loss
- Difficulty hearing

**Study Group 1 and Group 2 -** Possible side the usual radiation therapy used for this type of cancer:

#### **Possible Side Effects of Lung Radiation**

## **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving lung radiation, more than 20 and up to 100 may have:

- Swelling and redness, tanning, thickening, numbness, or peeling of the skin in the area of radiation
- Difficulty and/or pain with swallowing
- Hair loss in the treatment area, may be permanent
- Shortness of breath
- Cough with or without increased phlegm production
- Tiredness
- Anemia, which may require blood transfusion
- Infection, especially when white blood cell count is low
- Bleeding, bruising
- Rib pain, increased risk of rib fracture

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving lung radiation, from 4 to 20 may have:

- Inflammation of the lung that may cause difficulty breathing and can be life-threatening
- Narrowing of the throat which may cause vomiting, difficulty swallowing
- Scarring in the lung
- Lung collapse
- Fluid around lungs
- Bleeding from the lungs which may cause coughing up blood
- Fever
- Narrowing of the esophagus
- Pain in chest wall

#### RARE, AND SERIOUS

In 100 people receiving lung radiation, 3 or fewer may have:

- Abnormal opening in internal organs which may cause pain and bleeding
- Irritation of the heart causing heart failure, heart attack, chest pain, abnormal heartbeat, shortness of breath, swelling of ankles, cough or tiredness
- Transverse myelitis irritation of the spinal cord causing weakness, tingling or numbness of the lower body and legs, or paralysis of the lower half of the body
- Brachial plexopathy irritation of the nerves controlling the arm, causing weakness or paralysis
- Bleeding from the airway (windpipe)
- Narrowing of the airway causing shortness of breath
- Lung damage, may be life threatening
- Damage to the large blood vessels surrounding the heart, which could cause coughing up of blood and possibly death
- Sores and skin damage causing bleeding and severe pain and may lead to an open wound
- Death

**Study Group 2** - In addition to side effects listed above, people who are in Group 2 may also have some side effects from Atezolizumab (MPDL3280A). These side effects are listed below.

Risk Profile for Atezolizumab (MPDL3280A) (CAEPR Version 2.4, September 14, 2023)

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving atezolizumab (MPDL3280A), more than 20 and up to 100 may have:

- Tiredness
- Infection

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving atezolizumab (MPDL3280A), from 4 to 20 may have:

- Anemia which may require blood transfusion
- Diarrhea, nausea, vomiting
- Difficulty swallowing
- Fever
- Flu-like symptoms including body aches
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Reaction during or following a drug infusion which may cause fever, chills, rash
- Loss of appetite
- Pain in back
- Cough, shortness of breath, stuffy nose
- Itching, acne, rash

Atezolizumab (MPDL3280A) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Hormone gland problems (especially the thyroid, pituitary and adrenal glands, and pancreas). Signs and symptoms may include: headaches that will not go away or unusual headaches, extreme tiredness or changes in mood or behavior decreased sex drive; weight loss or weight gain; excessive thirst or urine; dizziness or fainting.
- Pain in belly
- Pain or swelling of the joints
- Rash that develops on skin, nails, scalp and inside of mouth or vagina that may be painful

#### RARE, AND SERIOUS

In 100 people receiving atezolizumab (MPDL3280A), 3 or fewer may have:

#### • Bruising, bleeding

Atezolizumab (MPDL3280A) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Heart problems including swelling and heart failure. Symptoms and signs of heart problems may include: shortness of breath, swelling of the ankles and body.
- A condition with high blood sugar which leads to tiredness, frequent urination or excessive thirst.
- Swelling and redness of the eye
- Intestinal problems (colitis) that can rarely lead to tears or holes in your intestine. Signs and symptoms of colitis may include: diarrhea or increase in bowel movements, blood in your stools or dark, tarry, sticky stools, severe belly pain or tenderness.
- Liver problems (hepatitis) which can cause liver failure. Signs and symptoms of hepatitis may include: yellowing of your skin or the whites of your eyes, severe nausea or vomiting; drowsiness; pain in the right upper belly.
- Damage to organs in the body when the body produces too many white cells
- Swelling of the brain (meningitis/encephalitis), which may cause: headache, confusion, sleepiness, seizures, and stiff neck.
- Abnormal movement of the facial muscles
- Swelling of the spinal cord
- Problem of the muscle, including swelling, which can cause muscle pain and severe muscle weakness sometimes with dark urine.
- Problem of the nerves that can cause paralysis. Signs and symptoms may include: numbness, tingling of hands and feet; weakness of the arms, legs.
- Kidney problems, including nephritis and kidney failure requiring dialysis. Signs of kidney problems may include: decrease in the amount of urine, blood in your urine, ankle swelling.
- Lung problems (pneumonitis and pleural effusion). Symptoms may include: new or worsening cough, chest pain, shortness of breath.
- Skin: blisters on the skin, including inside the mouth (can be severe), rash with blisters, skin rash developing 1-8 weeks after a drug is given, which may be accompanied by fever, lymph node swelling and organ failure.

#### **Additional Drug Risks**

The study drug may interact with other types of medications and herbal supplements. Your study doctor will give you a drug information that lists possible interactions. Share this information with your family members, caregivers, other health care providers, and pharmacists.

Rarely, there are problems getting enough supplies of the study drug. If that happens, your doctor will talk with you about your options.

## What are my responsibilities in this study? (03-NOV-2022)

If you choose to take part in this study you will need to:

- Keep your study appointments.
- Tell your doctor about:
  - o all medications and supplements you are taking because some medications and supplements may interact with the study drug
  - o any side effects
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study.

**For women:** Do not get pregnant or breastfeed while taking part in this study. **For men:** Do not father a baby while taking part in this study. **For all:** Tell your study doctor right away if you think that you or your partner have become pregnant during the study or within 5 months (150 days) after your last dose of study drug, atezolizumab.

## What are the costs of taking part in this study? (18-SEPT-2020)

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your small cell lung cancer. This includes:

- the costs of tests, exams, procedures, and drugs that you get during the study to monitor your safety, and prevent and treat side effects.
- the costs of getting the atezolizumab ready and giving it to you.
- your insurance co-pays and deductibles.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor or a member of the research team for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You and/or your insurance provider will not have to pay for exams, tests, and procedures done for research purposes only or that are covered by the study. These include:

• Submission of tumor tissue and blood for research.

You or your insurance provider will not have to pay for the atezolizumab while you take part in this study. The cost of getting the study drug ready and giving it to you is not paid by the study sponsor so you or your insurance company may have to pay for this. You will not have to pay

for hepatitis B/C testing, which is required if you have not been tested for hepatitis before entering the study.

Taking part in this study may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat your cancer. You may:

- Have more travel costs.
- Need to take more time off work.
- Have other additional personal costs.

You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment

## What happens if I am injured because I took part in this study?

If you are injured as a result of taking part in this study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in this study does not mean you give up these rights.

## Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

There are organizations that may look at your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group. Some of these organizations are:

- The study sponsor [NRG Oncology (NRG)]
- Any drug company supporting the study

- Other organizations in the National Clinical Trials Network (NCTN): Alliance for Clinical Trials in Oncology (ALLIANCE), ECOG-ACRIN Cancer Research Group (ECOG-ACRIN), SWOG, and Imaging and Radiation Oncology Core (IROC)
- The NCI Central IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The FDA and the groups it works with to review research, and similar ones if other countries are involved in the study.
- The NCI and the groups it works with to review research.
- The Cancer Trials Support Unit (CTSU), an organization sponsored by the NCI to provide greater access to cancer trials

Your study records also will be stored for future use. However, your name and other personal information will not be used. Some types of future research may include looking at your records and those of other patients to see who had side effects across many studies or comparing new study data with older study data. However, we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

## Where can I get more information? (01-OCT-2019)

You may visit the NCI web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

| You can talk to the study doctor about any questions or | concerns you have about this study or to |
|---|---|
| report side effects or injuries. Contact the study doctor | (insert |
| name of study doctor[s]) at | (insert telephone number). |
| For questions about your rights while in this study, call | the |
| (insert the name of organization or center) Institutional | Review Board at |
| (insert telephone num | aber). |

## Optional studies that you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. They are separate from the main study described above. These optional studies will not benefit your health. The researchers leading these optional studies hope the results will help other people

with your type of cancer in the future. The results will not be added to your medical records and you or your study doctor will not know the results.

Taking part in these optional studies is your choice. You can still take part in the main study even if you say "no" to any or all of these studies. There is no penalty for saying "no." You and your insurance company will not be billed for these optional studies. If you sign up for, but cannot complete any of these studies for any reason, you can still take part in the main study. Circle your choice of "yes" or "no" for each of the following studies.

# Optional sample collections for known laboratory studies and/or storage for possible future studies

Researchers are trying to learn more about cancer and other health problems using blood and tissue samples from people who take part in clinical trials. By studying these samples, researchers hope to find new ways to prevent, detect, treat, or cure diseases.

Some of these studies may be about how genes affect health and disease. Other studies may look at how genes affect a person's response to treatment. Genes carry information about traits that are found in you and your family. Examples of traits are the color of your eyes, having curly or straight hair, and certain health conditions that are passed down in families. Some of the studies may lead to new products, such as drugs or tests for diseases.

#### Known future studies

If you choose to take part in this optional study, researchers will collect blood for research on the genetic make-up of the blood cells, including sequencing of all or part of your DNA. This is called genomic sequencing. Sequencing allows researchers to identify your genetic code. Changes in your genetic code may be passed down through your family. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down. These are called germline changes.

#### **Unknown future studies**

If you choose to take part in these optional studies, blood and any remaining tumor tissue will be collected and stored. Storing samples for future studies is called "biobanking." The biobank is being run by NRG Oncology and is supported by the NCI. Also, any health-related information, such as your response to cancer treatment, results of study tests, and medicines you took, will be stored for future use. This is a publicly funded study. Samples from publicly funded studies are required to be shared as broadly as possible. However, we will protect your privacy. The goal of this is to make more research possible that may improve people's health.

The biobank is a public research resource. It has controlled access. This means that researchers who want to get samples and data from it must submit a specific research request. The request identifies who they are and what their planned research project is. Before getting the samples and data, the researchers must agree to keep the data private, only use it for their planned research project, and never use it to try to identify you.

We don't know what research may be done in the future using your blood samples. This means that:

- You will not be asked if you agree to take part in the future research studies.
- You and your study doctor will not be told when or what type of research will be done.
- Unknown future research studies also may include genomic sequencing of all or part of your DNA (as described above).
- You will not get reports or other information about any research that is done using your samples.

#### What is involved in this optional sample collection? (02-JUNE-2021)

If you agree to take part, here is what will happen next:

- 1. About 4 tablespoons of blood will be collected from a vein in your arm at the following time points: before you start treatment, at the end of treatment, and 3 months after CRT.
- 2. Samples from the tissue that was collected at the time your biopsy will be collected and sent to the biobank.
- 3. Your samples will be stored in the biobank. There is no limit on the length of time we will keep your samples and research information. The samples will be kept until they are used for research or destroyed.
- 4. Researchers can only get samples from the biobank after their research has been approved by experts.
- 5. Researchers will not be given your name or contact information.
- 6. Some of your genetic and health information may be placed in central databases for researchers to use. The databases will not include your name or contact information.

#### What are the risks in this optional sample collection?

- The most common risks related to drawing blood from your arm are brief pain and maybe a bruise.
- Generally, hospitals will keep some of your tissue. This tissue may be used to help treat your cancer in the future. There is a small risk that when this tissue sample is submitted to the biobank for this optional sample collection, your tissue could be used up.
- Your medical and genetic information is unique to you. There is a risk that someone
  outside of the research study could get access to your study records or trace information
  in a database back to you. They could use that information in a way that could harm you.
  Researchers believe the chance that someone could access and misuse your information is
  very small. However, the risk may increase in the future as people find new ways of
  tracing information.
- In some cases, this information could be used to make it harder for you to get or keep a job and get or keep health insurance. There are laws against the misuse of genetic information, but they may not give full protection. For more information about the laws that protect you, ask your study doctor or visit: https://www.genome.gov/10002328/.

#### How will information about me be kept private?

Your privacy is very important to the study researchers and biobank. They will make every effort to protect it. Here are just a few of the steps they will take:

- 1. They will remove identifiers, such as your initials, from your sample and information. They will replace them with a code number. There will be a master list linking the code numbers to names, but they will keep it separate from the samples and information.
- 2. Researchers who study your sample and information will not know who you are. They also must agree that they will not try to find out who you are.
- 3. Your personal information will not be given to anyone unless it is required by law.
- 4. If research results are published, your name and other personal information will not be used.

#### What are the benefits to taking part in this optional sample collection?

You will not benefit from taking part.

The researchers, using the samples from you and others, might make discoveries that could help people in the future.

## Are there any costs or payments to this optional sample collection?

There are no costs to you or your insurance. You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

| any payment. |
|---|
| What if I change my mind about this optional sample collection? If you decide you no longer want your samples to be used, you can call the study doctor, |
| let the biobank know. Then, any sample that remains in the biobank will be destroyed or returned to your study doctor. This will not apply to any samples or related health information that have already been given to or used by researchers. |
| What if I have questions about this optional sample collection? If you have questions about the use of your samples for research, contact the study doctor, |
| (insert telephone number of study doctor for main trial). |
| Please circle your answer below to show if you would or would not like to take part in each optional study: |
| Samples for known future studies: I agree that my samples and related health information may be used for the laboratory studies described above. |
| YES NO |

#### Samples for unknown future studies:

I agree that my samples and related health information may be kept in a biobank for use in future health research.

YES NO

#### **Contact for Future Research**

I agree that my study doctor, or someone on the study team, may contact me or my doctor to see if I wish to participate in other research in the future.

YES NO

This is the end of the section about optional studies.

## My signature agreeing to take part in the study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed and dated copy of this form. I agree to take part in the main study. I also agree to take part in any additional studies where I circled "yes".

| Participant's signature |
|-------------------------------------------------------------------|
| Date of signature |
| Success Signature |
| Signature of person(s) conducting the informed consent discussion |
| Date of signature |

## **Appendix I: Patient Instructions for Accessing the Patient Cloud Using Your Personal Device (01-OCT-2019)**

Downloading the Patient Cloud ePRO App

If you are using your personal device, and you do not have the Patient Cloud ePRO app, use the following instructions. When downloading the app, you must use the Apple ID or Google account associated with the device. If the Patient Cloud ePRO app is already on the device, or if you are using a provider's device, you can skip this section.

You will need an email address that you agree to use for this purpose. The e-mail address is needed to identify you on the Patient Cloud Application and for you to receive notifications to let you know when forms are due. Your e-mail address will only be used for this survey study, and will not be used for mail or marketing purposes.

If you decide to use the electronic method to complete the questionnaires, and do not have an email address, you may sign up for one at no charge at many different websites. A few sites that are commonly used and will allow you to create an email address very easily are <u>Yahoo</u>, <u>Gmail</u>, and <u>Outlook</u>.

#### For iOS:

- 1. An Apple ID is required for downloading the Patient Cloud ePRO app.
- 2. Tap the *App Store* icon.
- 3. Search for *Medidata Patient Cloud* and follow the installation instructions.

Note: Patient Cloud ePRO is listed as an iPhone App in the App store. When using an iPad, please view the search results under iPhone apps.

#### For Android:

- 1. A Google account is required for downloading the Patient Cloud ePRO app
- 2. Tap the *Play Store* icon.
- 3. Search for *Medidata Patient Cloud* and follow the installation instructions.

#### Registering

You must register in order to complete and submit your study forms. When you register, you will create a username, which is your email address, and a password that allows you to log in to the Patient Cloud ePRO app.

Note: You must have an activation code to begin this process. If you do not have an activation code, please contact your provider.

There are two possible ways to register. Your provider may have sent you a link to a web address where you may register from any web browser, including the one on your device. The other way to register is on the Patient Cloud ePRO app.

- 1. If registering from the Patient Cloud app, tap Register on the bottom of the log in page. If registering on the web, open the URL shield.imedidata.com on a web browser.
- 2. Enter your activation code and tap Activate.
- 3. On the next page, read the instructions and tap Next.
- 4. Read the privacy notice and tap I agree. Then tap OK to confirm.
- 5. Enter and confirm your email address. Tap Next.
- 6. Enter and confirm your password. Tap Next.
- 7. Choose a security question by scrolling through the dropdown menu to display the question of your choice.
- 8. Enter your security question response.
- 9. Tap Create my account to complete your registration.

If you registered on the Patient Cloud ePRO app, it automatically logs you out. If you registered on the web, you are presented with the option to download the Patient Cloud ePRO app. You can then proceed to log in with the credentials you created.

#### Logging in to the App

- 1. Enter your Email and Password that you created during the registration process. (If you previously set a PIN code, just enter your four-digit PIN.)
- 2. Tap Log in.

Note: If you do not remember your password, tap **Forgot Password**, and follow the instructions provided.

#### Setting a PIN Code

The first time you log in to the Patient Cloud ePRO app, you are given the option to create a PIN code. A PIN code allows you to bypass the step of entering your email and password every time you need to log in to the Patient Cloud ePRO app. Instead, you can enter a four-digit PIN.

- 1. If you wish to set a PIN code the first time you log in, tap Yes when prompted.
- 2. Note: You can also set your PIN at a later time by tapping the options menu on the top left of most pages and selecting Set PIN.
- 3. Enter a four-digit PIN.
- 4. Re-enter the four-digit PIN to confirm.

If you forget your PIN code, tap **Forgot PIN** and you can access the app using your email and password. You may reset your PIN by tapping the options menu on the top left of most pages and selecting Set PIN.

#### Resetting Your Password

You can reset your password by using the options menu at the top left of most pages.

- 1. Tap the options menu icon.
- 2. Tap Reset Password.
- 3. Follow the instructions to reset your password.

#### Completing and Submitting Forms

Once logged in, forms related to your study display on the Tasks page. If you are enrolled in multiple studies, select the appropriate study first, and then select a form. New forms can appear on the Tasks page at any time, depending on how the study is designed.

There are two types of forms displayed on the Task List page:

- Scheduled Forms (with a icon): These forms have a "Due Date" indicator in them so you are aware of the last day by which you will need to complete the form. If the form is due in less than one day, you will see the due time in hours.
- Anytime Forms (with a icon): These forms have "Last Completed Time" indicator on them which tells the most recent date or time when you completed the form. If you start a form, but do not complete it, you will see an 'Incomplete" status beneath the form name, along with a half-moon icon.
  - 1. Select the appropriate form.
  - 2. Follow the on-screen instructions until you reach the end of the form where you are given the opportunity to review and change your responses prior to submitting.
  - 3. Review your responses by scrolling down the list.
  - 4. If you need to change an answer, tap the question to go back and change the answer.
  - 5. When you are ready to submit, tap Submit Your Data.

Note: Once a form is submitted, you will be unable to edit any of your responses. In some cases, you may be asked to acknowledge your submission by entering your password.